CLINICAL TRIAL: NCT00626327
Title: A Phase 3, Open-Label, Randomized, Multi-Center Study to Evaluate the Safety and Immunogenicity of MMRV Vaccine When Administered Concomitantly With Novartis Meningococcal ACWY Conjugate Vaccine to Healthy Toddlers
Brief Title: Safety and Immune Response of Novartis MenACWY-CRM Conjugate Vaccine When Given to Healthy Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V59P21; BB-IND 11278
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Results first posted 2013-03-15 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Meningococcal Infections
Keywords: vaccine; toddlers; healthy; meningitis; meningococcal; measles; mumps; rubella; varicella; Prevention of Meningococcal disease types ACWY
MeSH Terms: conditions — Meningococcal Infections; Meningitis; Measles; Mumps; Rubella; Chickenpox | interventions — measles, mumps, rubella, varicella vaccine; MenACWY-CRM vaccine

ARMS (3):
- MenACWY-CRM+ MMRV (Experimental)
  Interventions: Biological: MenACWY-CRM + MMRV
- MMRV (Active Comparator)
  Interventions: Biological: MMRV
- MenACWY-CRM (Experimental)
  Interventions: Biological: MenACWY-CRM

INTERVENTIONS:
Biological: MenACWY-CRM + MMRV — One injection of MenACWY-CRM vaccine at 7-9 months of age; the second injection of MenACWY-CRM vaccine concomitantly administered with MMRV (Measles, Mumps, Rubella and Varicella) vaccine at 12 months of age.
  Arms: MenACWY-CRM+ MMRV
Biological: MMRV — one injection of MMRV (Measles, Mumps, Rubella and Varicella) vaccine at 12 months of age
  Arms: MMRV
Biological: MenACWY-CRM — Two injections of MenACWY-CRM at 7-9 months and 12 months of age; one injection of MMRV (Measles, Mumps, Rubella and Varicella) at 13.5 months of age
  Arms: MenACWY-CRM

SUMMARY:
Safety immune response of Novartis MenACWY-CRM conjugate vaccine when given to healthy toddlers

ELIGIBILITY:
Inclusion Criteria:

* who are healthy 7 to 9 months old or 12 months old (inclusive plus 14 days) and for whom, after the nature of the study has been explained, the parent or legal guardian has provided written informed consent;
* who have received complete primary vaccination with recommended licensed vaccines;
* who are available for all visits and telephone calls scheduled for the study;

Exclusion Criteria:

* whose parent or legal guardian is unwilling or unable to give written informed assent consent
* who had a previous or suspected disease caused by N. meningitidis;
* who had previous or suspected infection with measles, mumps, rubella, varicella, and/or herpes zoster;
* who had household contact with and/or intimate exposure to an individual with culture-proven N. meningitidis infection within 60 days prior to enrollment;
* who had household contact with and/or intimate exposure to an individual with measles, mumps, rubella and/or varicella infection within 60 days prior to enrollment;
* who have previously been immunized with a meningococcal vaccine or vaccine containing meningococcal antigen(s)
* who have previously received any measles, mumps, rubella or varicella vaccine either alone or in any combination;
* who have received any investigational agents or vaccines within 90 days prior to enrollment or who expect to receive an investigational agent or vaccine prior to the completion of the study;
* who have any serious acute, chronic or progressive disease such as, cancer, diabetes, heart failure, malnutrition, epilepsy, HIV/AIDS, Guillain Barre Syndrome
* who have a history of anaphylaxis, serious vaccine reactions or allergy to any part of the vaccine,
* who have a known or suspected impairment/alteration of immune function, either congenital or acquired
* who have Down's syndrome or other known cytogenic disorders; bleeding diathesis

Ages: 7 Months to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1630 (Actual)
Dates: Start 2008-02; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (90):
- United States (90):
  - Site 85 - Birmingham Pediatric Associates, 806 St. Vincent's Drive, Birmingham, Alabama
  - Site 86 - Southeastern Pediatrics Associate, 364 Honeysuckle Road, Dothan, Alabama
  - Site 00 - Veritas Research LLC/ Stabler Clinic, 300 North College Street,, Greenville, Alabama
  - Site 42 - Drug Research and Analysis Corporation, 1758 Parkplace, Suite 200, Montgomery, Alabama
  - Site 56 - Children's Investigational Research Program, LLC, 2719 SE I Street, Bentonville, Arkansas
  - Site 94 - Central Arkansas Pediatrics, 2425 Dave Ward Dr.; Suite 601, Conway, Arkansas
  - Site 80 - The Children's Clinic of Jonesboro, 800 S. Church St; Suite 400; 4th Fl, Jonesboro, Arkansas
  - Site 49 - Arkansas Pediatric Clinical Research, 500 S. University; Suite 200, Little Rock, Arkansas
  - Site 05 - Kaiser Permanente Pediatric Clinic 395 Hickory Blvd. 2nd Floor; Room 265, Daly City, California
  - Site 08 - Kaiser Permanente Pediatric Clinic 4785 N. First Street 3rd Floor, Fresno, California
  - Site 70 - Loma Linda University, Department of Pediatrics, 11175 Campus Street; CP A1120, Loma Linda, California
  - Site 71 - LLUHC Moreno Valley Pediatrics, 11401 Heacock Street, Moreno Valley, California
  - Site 34 - Children's Hospital and Research Center Oakland (CHRCO), Infectious Diseases Department, 747 52nd Street, Oakland, California
  - Site 72 - Children's Hospital of Orange Co. 455 South Main Street, Orange, California
  - Site 58 - Center for Clinical Trials, LLC 16660 Paramount Boulevard Suite 301, Paramount, California
  - Site 59 - Center for Clinical Trials, LLC 16415 S. Colorado Avevue Suite 308, Paramount, California
  - Site 04 - Kaiser Permanente Pediatric Clinic, 610 Walnut Street, Room 110, Redwood City, California
  - Site 37 - Kaiser Permanente Pediatric Clinic 901 Nevin Ave. Room 1E24, Richmond, California
  - Site 09 - Kaiser Permanente Pediatric Clinic 1840 Sierra Gardens Vaccine Studies, Roseville, California
  - Site 03 - Kaiser Permanente Pediatric Clinic, Point West Medical Offices, 1650 Response Road, Sacramento, California
  - Site 48 - Pediatric Infectious Diseases Admin 2516 Stockton Blvd.; Ticon II, Sacramento, California
  - Site 10 - Kaiser Permanente Pediatric Clinic 6600 Bruceville Road Pediatric Station C, Sacramento, California
  - Site 50 - Kaiser Permanente Pediatric Clinic 3925 Old Redwood Hwy, Santa Rosa, California
  - Site 24 - UCLA Center for Vaccine Research 1124 W Carson St., Torrance, California
  - Site 07 - Kaiser Permanente Pediatric Clinic 975 Sereno Drive; 1st Floor MOB Pediatric Station 1, Vallejo, California
  - Site 02 - Kaiser Permanente Pediatric Clinic, 1425 S. Main Street; MOB2, 4th Floor; Station 2, Walnut Creek, California
  - Site 40 - 1st Allergy and Asthma Center 3260 E. 104th Ave.; Suite C, Thornton, Colorado
  - Site 41 - 1st Immunology & Clinical Research 3260 East 104th Avenue, Thornton, Colorado
  - Site 60 - Norwich Pediatric Group, PC 92 New London Turnpike, Norwich, Connecticut
  - Site 47 - Department of Clinical Trials 1401Lucerne Terrace; MP141, Orlando, Florida
  - Site 25 - Kentucky Pediatric/ Adult Research 201 South 5th Street Suite 102, Bardstown, Kentucky
  - Site 52 - Cincinnati Children's Hosp Med Ctr Gamble Program for Clinical Studies 2865 Chancellor Drive, Crestview Hills, Kentucky
  - Site 74 - University of Louisville University Child Health Specialists 230 East Broadway, Louisville, Kentucky
  - Site 87 - University of Louisville Children & Youth Project 555 South Floyd Street, Louisville, Kentucky
  - Site 88 - University of Louisville Univ. of Child Health Specialist So 9702 Stonestreet Road; Suite 100, Louisville, Kentucky
  - Site 57 - Bluegrass Clinical Research, Inc. 5512 Bardstown Rd; Suite 2, Louisville, Kentucky
  - Site 84 - Springs Medical Research, PLLC 2200 East Parrish Avenue Suite 101, Owensboro, Kentucky
  - Site 68 - Physicians to Children/ Adolescents 102 West Depot Street, Springfield, Kentucky
  - Site 93 - ACC Pediatric Research 1025 Highway 80 East, East Haughton, Louisiana
  - Site 63 - Ochsner Clinic Foundations, 1315 Jefferson Highway, New Orleans, Louisiana
  - Site 39 - Pediatric Associates of Fall River, 829 S. Main Street, Fall River, Massachusetts
  - Site 96 - Southwestern Medical Clinic, PC 2002 South 11th Street, Niles, Michigan
  - Site 89 - Southwestern Medical Clinic 5515 Cleveland Ave.; Suite 1, Stevensville, Michigan
  - Site 73 - University of MS Medical Ctr Pediatric Clinical Research 2500 North State St; 2 East-H255, Jackson, Mississippi
  - Site 79 - Children's Physicians Bellevue 11507 S. 42nd Street, Bellevue, Nebraska
  - Site 66 - Creighton University Department of Pediatrics 601 N. 30th St.; Suite 6820, Omaha, Nebraska
  - Site 78 - Children's Physicians Dundee 119 North 51st Street, Omaha, Nebraska
  - Site 76 - Winthrop University Hospital Winthrop Pediatric Associates 120 Mineola Boulevard, Suite 210, Mineola, New York
  - Site 91 - SUNY Upstate Medical University 750 East Adams St,; Suite 5400, Syracuse, New York
  - Site 77 - Montefiore Medical Center 111 East 210th Street Rosenthall Building; 4th Floor, The Bronx, New York
  - Site 28 - Duke Health Center at Roxboro Road 4020 North Roxboro Road, Durham, North Carolina
  - Site 29 - Regional Pediatrics 4022 Freedom Lake Drive, Durham, North Carolina
  - Site 30 - Durham Pediatrics 2609 North Duke Street Suite 100, Durham, North Carolina
  - Site 82 - Austintown Pediatrics 107 Javit Court, Austintown, Ohio
  - Site 51 - Cincinnati Children's Hosp Med Ctr Gamble Program for Clinical Studies 3333 Burnet Avenue; MLC 6014, Cincinnati, Ohio
  - Site 62 - Dr. Senders and Assoc., Pediatrics 2054 South Green Road, Cleveland, Ohio
  - Site 97 - Dayton Clinical Research 1100 Salem Avenue, Dayton, Ohio
  - Site 35 - Caro Pediatric Center 111 Turner Road, Dayton, Ohio
  - Site 26 - Ohio Pediatrics 7371 Brandt Pike; Suite C, Huber Heights, Ohio
  - Site 27 - Ohio Pediatrics 1775 Delco Park Drive, Kettering, Ohio
  - Site 90 - OK State Univ-Ctr for Health Scienc Houston Parke Physicians 635 W. 11th StreetOklahoma State University - Center for Health Sciences, Tulsa, Oklahoma
  - Site 31 - Calcagno Research and Development 24850 SE Stark Street Suite 150, Gresham, Oregon
  - Site 32 - Drexel Hill Pediatrics 5030 State Rd.; Suite 2-900, Drexel Hill, Pennsylvania
  - Site 13 - Children's Health Care- West 4671 West Lake Road, Erie, Pennsylvania
  - Site 15 - UPMC/ Community Medicine, Inc 90 Shenango Street, Greenville, Pennsylvania
  - Site 19 - Pediatric Associates of Latrobe 210 Welson Street, Latrobe, Pennsylvania
  - Site 18 - Squirrel Hill Office 4070 Beechwood Blvd, Pittsburgh, Pennsylvania
  - Site 21 - Pediatric Alliance Greentree Div. 969 Greentree Road Suite 100, Pittsburgh, Pennsylvania
  - Site 20 - South Hill Pediatrics 4411 Stilley Road, Pittsburgh, Pennsylvania
  - Site 17 - Pediatric Alliance, Southwestern, 850 Clairton Blvd, Pittsburgh, Pennsylvania
  - Site 83 - Pediatric Alliance, PC Arcadia Division 9000 Perry Hwy; Suite 120, Pittsburgh, Pennsylvania
  - Site 12 - Pediatric Alliance St. Clair 1580 McLaughlin Run Road, Pittsburgh, Pennsylvania
  - Site 16 - Laurel Pediatrics 140 Wayland Smith Drive, Uniontown, Pennsylvania
  - Site 14 - CCP - Pittsburgh Pediatrics 6000 Brooktree Road Suite 207, Wexford, Pennsylvania
  - Site 81 - Alpha Clinical Research, LLC 279 Clear Sky Court; Suite C, Clarksville, Tennessee
  - Site 11 - Focus Research Group 242 West Main, Hendersonville, Tennessee
  - Site 38 - Jackson Clinic 2683 Highway 45 Bypass North, Jackson, Tennessee
  - Site 69 - University of North Texas Health Science Center 855 Montgomery Street, Fort Worth, Texas
  - Site 36 - Pediatric Healthcare of Northwest Houston P.A. 13406 Medical Complex Drive Suite 200, Houston, Texas
  - Site 43 - Wee Care Pediatrics 1580 W. Antelope Drive; Suite 100, Layton, Utah
  - Site 45 - Wee Care Pediatrics 934 South Main St.; Suite 8, Layton, Utah
  - Site 44 - Wee Care Pediatrics 5991 South 3500 West; Suite 100 Rock Run Plaza, Roy, Utah
  - Site 53 - Copperview Medical Center 3556 West 9800 South Suite 101, South Jordan, Utah
  - Site 67 - Virginia Commonwealth Univ. 1001 East Marshall Street Room P008, Richmond, Virginia
  - Site 55 - Children's Hosp. & Regional Med Ctr 4800 Sand Point Way NE; MS 5441, Seattle, Washington
  - Site 06 - Rockwood Clinic, P.S. 400 East Fifth Avenue, Spokane, Washington
  - Site 46 - Rockwood Clinic North 9001 N. Country Homes Blvd, Spokane, Washington
  - Site 98 - University Physicians Internal Medicine 1600 Medical Center Drive, Huntington, West Virginia
  - Site 92 - Gundersen Clinic, Ltd. 1836 South Ave.; Mailstop C03-006B, La Crosse, Wisconsin
  - Site 64 - Monroe Medical Foundation Monroe Clinic 515 22nd Avenue, Monroe, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 90 centers in the USA
Pre-assignment Details: All subjects enrolled were included in the trial.
Groups:
- MenACWY-CRM+ MMRV: Subjects in this group received 2 injections of MenACWY-CRM at 7-9 and 12 months; second injection administered concomitantly with MMRV
- MMRV: Subjects in this group received 1 injection of MMRV vaccine at 12 months of age
- MenACWY-CRM: Subjects in this group received 2 injections of the MenACWY-CRM vaccine at 7-9 and 12 months of age followed by 1 injection of MMRV at 13.5 months
Period: Overall Study
Arm/Group | MenACWY-CRM+ MMRV | MMRV | MenACWY-CRM
Started | 504 | 616 | 510
Completed | 426 | 557 | 422
Not Completed | 78 | 59 | 88
Not completed — Withdrawal by Subject | 21 | 29 | 30
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 24 | 21 | 23
Not completed — Inappropriate enrollment | 4 | 5 | 3
Not completed — Administrative Reason | 2 | 0 | 6
Not completed — Protocol Violation | 26 | 4 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MenACWY-CRM+ MMRV | MMRV | MenACWY-CRM | Total
Number analyzed (Participants) | 504 | 616 | 510 | 1630
Age Continuous [Mean (Standard Deviation); unit: months] | 8.5 (0.8) | 12.1 (0.3) | 8.5 (0.8) | 9.8 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 251 | 304 | 252 | 807
  Male | 253 | 312 | 258 | 823

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With a Seroresponse to Measles, Mumps, Rubella and Varicella Following Concomitant Administration of MMRV Vaccine With MenACWY-CRM Vaccine
Description: Percentages of subjects with seroresponses to measles, mumps, rubella and varicella after one dose of MMRV vaccine (at 12 months) when given concomitantly with MenACWY-CRM vaccine compared to when MMRV vaccine was given alone, are reported.
  Seroresponse was defined as the percentage of initially seronegative subjects who show seroconversion to measles (≥255 mIU/mL), mumps (≥10 ELISA Ab units), rubella (≥10 IU/mL) and the percentage of initially seronegative subjects who show seroprotection (≥5 gp ELISA units/mL) for varicella.
  Immunogenicity to measles, mumps, rubella and varicella at 6 weeks after vaccination with one dose of MMRV given concomitantly with MenACWY-CRM was considered non-inferior to immunogenicity of MMRV administered alone if the lower limit of two-sided 95% CI of the difference in the percentage of subjects with seroconversion for measles, mumps, and rubella, and seroprotection for varicella was greater than -5% (measles, mumps and rubella) and -10% (varicella).
Time Frame: 6 weeks post vaccination
Population: The analysis was performed on the MMRV per-protocol population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY-CRM+ MMRV | MMRV
Number analyzed (Participants) | 370 | 515
Percentages of subjects
  Measles (N=350,467) | 98 [96 to 99] | 99 [98 to 100]
  Mumps (N=365,499) | 98 [96 to 99] | 96 [94 to 98]
  Rubella | 95 [93 to 97] | 97 [95 to 98]
  Varicella (N=337,459) | 96 [94 to 98] | 98 [96 to 99]
Statistical Analysis 1: Comparison: MenACWY-CRM+ MMRV vs MMRV; Non-inferiority of immune response to measles following one dose of MMRV administered concomitantly with MenACWY-CRM as compared to MMRV given alone; Test type: Non-Inferiority or Equivalence — The immune response of MenACWY-CRM+MMRV group was considered non-inferior to that of MMRV group if the lower limit of the two-sided 95% CI of the difference in the percentage of subjects with seroconversion for measles was greater than -5%, at 6 weeks after MMRV vaccination; Difference % (MenACWY-CRM+MMRV-MMRV) = -1, 95% CI 2-sided [-3.4 to 0.5]
Statistical Analysis 2: Comparison: MenACWY-CRM+ MMRV vs MMRV; Non-inferiority of immune response to mumps following one dose of MMRV administered concomitantly with MenACWY-CRM as compared to MMRV administered alone; Test type: Non-Inferiority or Equivalence — The immune response of MenACWY-CRM+MMRV group was considered non-inferior to that of MMRV group if the lower limit of the two-sided 95% CI of the difference in the percentage of subjects with seroconversion for mumps was greater than -5%, at 6 weeks after MMRV vaccination; Difference % (MenACWY-CRM+MMRV - MMRV ) = 1, 95% CI 2-sided [-1 to 3.7]
Statistical Analysis 3: Comparison: MenACWY-CRM+ MMRV vs MMRV; Non-inferiority of immune response to rubella following one dose of MMRV administered concomitantly with MenACWY-CRM as compared to MMRV administered alone; Test type: Non-Inferiority or Equivalence — The immune response of MenACWY-CRM+MMRV group was considered non-inferior to that of MMRV group if the lower limit of the two-sided 95% CI of the difference in the percentage of subjects with seroconversion for rubella was greater than -5%, at 6 weeks after MMRV vaccination; Difference% (MenACWY-CRM+MMRV-MMRV) = -2, 95% CI 2-sided [-4.5 to 0.8]
Statistical Analysis 4: Comparison: MenACWY-CRM+ MMRV vs MMRV; Non-inferiority of immune response to varicella following one dose of MMRV administered concomitantly with MenACWY-CRM as compared to MMRV administered alone; Test type: Non-Inferiority or Equivalence — The immune response of MenACWY-CRM+MMRV group was considered non-inferior to that of MMRV group if the lower limit of the two-sided 95% CI of the difference in the percentage of subjects with seroprotection for varicella was greater than -10%, at 6 weeks after MMRV vaccination; Difference% (MenACWY-CRM+MMRV-MMRV) = -1, 95% CI 2-sided [-3.9 to 1.2]

2. Primary Outcome: Percentages of Subjects With Serum Bactericidal Titers ≥1:8 Following Concomitant Administration of MenACWY-CRM Vaccine With MMRV Vaccine.
Description: Percentages of subjects with hSBA ≥1:8, against N.meningitidis serogroups A, C, W-135, and Y following two doses of MenACWY-CRM vaccine (at 7-9 months and 12 months) when concomitantly administered with MMRV vaccine (12 months) compared to when MenACWY-CRM vaccine was given alone, are reported.
  The serum bactericidal antibodies directed against N.meningitidis serogroups A, C, W-135, and Y, were measured by human complement Serum Bactericidal Assay (hSBA).
  The immune response of MenACWY-CRM given concomitantly with MMRV was considered non-inferior to the immunogenicity of MenACWY-CRM administered alone if the lower limit of the two-sided 95% CI around the difference of the percentage of subjects with hSBA ≥1:8 at 6 weeks after the second dose of MenACWY-CRM given to 12-month old toddlers {P MMRV+MenACWY minus P MenACWY} was greater than -10% for each serogroup.
Time Frame: 6 weeks post second dose
Population: The analysis was performed on the MenACWY per-protocol population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY-CRM+ MMRV | MenACWY-CRM
Number analyzed (Participants) | 384 | 379
Percentages of subjects
  Serogroup A | 88 [84 to 91] | 88 [84 to 91]
  Seroroup C (N=204,195) | 100 [98 to 100] | 100 [98 to 100]
  Sergroup W-135 (N=204,196) | 100 [97 to 100] | 98 [96 to 100]
  Serogroup Y (N=200,198) | 98 [95 to 99] | 96 [93 to 99]
Statistical Analysis 1: Comparison: MenACWY-CRM+ MMRV vs MenACWY-CRM; Non-inferiority of immune response of MenACWY-CRM against serogroup A when concomitantly administered with MMRV vaccine as compared to MenACWY-CRM vaccine given alone; Test type: Non-Inferiority or Equivalence — The immune response of MenACWY-CRM + MMRV group was considered non-inferior to that of MenACWY-CRM group if the lower limit of the two-sided 95% CI around the difference of the percentage of subjects with hSBA ≥1:8 at 6 weeks after the second dose of MenACWY-CRM given to 12 month old toddlers was greater than -10% for each serogroup; Difference% (MenACWY-CRM+MMRV-MenACWY) = 0, 95% CI 2-sided [-4.7 to 4.5]
Statistical Analysis 2: Comparison: MenACWY-CRM+ MMRV vs MenACWY-CRM; Non-inferiority of immune response of MenACWY-CRM against serogroup C when concomitantly administered with MMRV vaccine as compared to MenACWY-CRM vaccine given alone; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference% (MenACWY-CRM+MMRV-MenACWY) = 0, 95% CI 2-sided [-1.8 to 1.9]
Statistical Analysis 3: Comparison: MenACWY-CRM+ MMRV vs MenACWY-CRM; Non-inferiority of immune response of MenACWY-CRM against serogroup W-135 when concomitantly administered with MMRV vaccine as compared to MenACWY vaccine given alone; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference% (MenACWY-CRM+MMRV-MenACWY) = 1, 95% CI 2-sided [-1.3 to 3.9]
Statistical Analysis 4: Comparison: MenACWY-CRM+ MMRV vs MenACWY-CRM; Non-inferiority of immune response of MenACWY-CRM against serogroup Y when concomitantly administered with MMRV vaccine as compared to MenACWY-CRM vaccine given alone; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference% (MenACWY-CRM+MMRV-MenACWY) = 2, 95% CI 2-sided [-1.9 to 5.3]

3. Primary Outcome: Percentages of Subjects With hSBA ≥1:8 Following Two Doses of MenACWY-CRM Vaccine
Description: The antibody response following two doses of MenACWY-CRM vaccine (at 7-9 months and 12 months) was considered adequate if the lower limit of the two-sided 95% CI for the percentage of subjects with hSBA ≥1:8, at 6 weeks following the second dose of MenACWY-CRM, was greater than 85% for serogroups C, W-135, or Y and greater than 65% for serogroup A.
Time Frame: 6 weeks post vaccine dose 2
Population: The analysis was performed on the MenACWY per-protocol population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY-CRM
Number analyzed (Participants) | 379
Percentages of subjects
  Serogroup A | 88 [84 to 91]
  Serogroup C (N=195) | 100 [98 to 100]
  Serogroup W-135 (N=196) | 98 [96 to 100]
  Serogroup Y (N=198) | 96 [93 to 99]

4. Secondary Outcome: Percentages of Subjects With hSBA ≥1:4 After Two Doses of MenACWY-CRM Vaccine
Description: The percentages of subjects with hSBA ≥1:4 directed against N. meningitidis serogroups A, C, W-135, and Y following two doses of MenACWY-CRM vaccine (at 7-9 and 12 months of age) when given concomitantly with MMRV vaccine (at 12 months) compared to when MenACWY-CRM vaccine was given alone, are reported.
Time Frame: 6 weeks post vaccine dose 2
Population: The analysis was performed on the MenACWY per-protocol population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- MenACWY-CRM+MMRV: Subjects in this group received 2 injections of MenACWY-CRM at 7-9 and 12 months; second injection administered concomitantly with MMRV
Arm/Group | MenACWY-CRM+MMRV | MenACWY-CRM
Number analyzed (Participants) | 384 | 379
Percentages of subjects
  Serogroup A | 90 [86 to 92] | 91 [87 to 93]
  Serogroup C (N=204,195) | 100 [98 to 100] | 100 [98 to 100]
  Serogroup W-135 (N=204,196) | 100 [97 to 100] | 99 [96 to 100]
  Serogroup Y (N=200,198) | 98 [95 to 99] | 98 [95 to 99]

5. Secondary Outcome: Geometric Mean Titers Against Serogroups A, C, W-135 and Y, Following Two Doses of MenACWY-CRM Vaccine
Description: The geometric mean titers (GMTs) directed against N.meningitidis serogroups A, C, W-135 and Y, following two doses of MenACWY-CRM vaccine (at 7-9 months and 12 months of age), when given concomitantly with MMRV vaccine (at 12 months) compared to when MenACWY-CRM vaccine was given alone, are reported.
Time Frame: 6 weeks post vaccine dose 2
Population: The analysis was performed on the MenACWY per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- MenACWY-CRM + MMRV: Subjects in this group received 2 injections of MenACWY-CRM at 7-9 and 12 months; second injection administered concomitantly with MMRV
Arm/Group | MenACWY-CRM + MMRV | MenACWY-CRM
Number analyzed (Participants) | 384 | 379
Titers
  Serogroup A | 39 [34 to 45] | 37 [32 to 42]
  Serogroup C (N=204,195) | 194 [170 to 220] | 180 [158 to 205]
  Serogroup W-135 (N=204,196) | 132 [113 to 155] | 119 [101 to 139]
  Serogroup Y (N=200,198) | 97 [81 to 116] | 88 [73 to 105]

6. Secondary Outcome: Geometric Mean Titers Against Measles, Mumps, Rubella and Varicella Following One Dose of MMRV Vaccine.
Description: The GMTs directed against measles, mumps, rubella and varicella, following one dose of MMRV vaccine (at 12 months) when given concomitantly with MenACWY-CRM vaccine compared to when MMRV vaccine was given alone, are reported.
Time Frame: 6 weeks post vaccination
Population: The analysis was performed on the MMRV per-protocol population.
  Only subjects with a baseline titer below the specified cut-off for that antigen were included in the immunogenicity analysis for the same antigen.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM+ MMRV | MMRV
Number analyzed (Participants) | 377 | 518
Titers
  Pre-dose, Measles (N=357,470) | 74 [71 to 77] | 74 [71 to 77]
  Post-dose, Measles (N=350,467) | 4049 [3701 to 4430] | 3632 [3350 to 3938]
  Pre-dose, Mumps (N=372,502) | 5 [5 to 5] | 5 [5 to 5]
  Post-dose, Mumps (N=365,499) | 97 [89 to 107] | 81 [75 to 88]
  Pre-dose, Rubella | 5 [5 to 5] | 5 [5 to 5]
  Post-dose, Rubella (N=370,515) | 57 [52 to 62] | 56 [52 to 61]
  Pre-dose, Varicella (N=344,461) | 0.63 [0.63 to 0.63] | 0.63 [0.63 to 0.63]
  Post-dose, Varicella (N=337,459) | 19 [17 to 20] | 18 [17 to 19]

7. Secondary Outcome: Percentages of Subjects Showing Seroconversion Response to Varicella Following Concomitant Administration of MMRV With MenACWY-CRM Vaccine.
Description: The percentages of subjects showing seroconversion response to varicella after concomitant administration of MMRV vaccine (at 12 months) with MenACWY-CRM vaccine compared to when MMRV vaccine is given alone, is reported .
  Seroconversion for varicella is defined as percentage of subjects who show pre-vaccination antibody titer <1.25 gp ELISA units/mL to a post-vaccination antibody titer ≥1.25 gp ELISA units/mL.
Time Frame: 6 weeks post vaccination
Population: The analysis was performed on the MMRV per-protocol population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- MenACWY-CRM +MMRV: Subjects in this group received 2 injections of MenACWY-CRM at 7-9 and 12 months; second injection administered concomitantly with MMRV
Arm/Group | MenACWY-CRM +MMRV | MMRV
Number analyzed (Participants) | 337 | 459
Percentages of subjects | 99 [97 to 100] | 99 [98 to 100]
Statistical Analysis 1: Comparison: MenACWY-CRM +MMRV vs MMRV; Non-inferiority of anti-varicella response following one dose of MMRV when administered concomitantly with MenACWY vaccine as compared to MMRV administered alone; Test type: Non-Inferiority or Equivalence — The immune response of MMRV+MenACWY group was considered non-inferior to that of MMRV group if the lower limit of the two-sided 95% CI of the difference in the percentages of subjects with seroconversion for varicella was greater than -10%; Difference% (MenACWY-CRM+MMRV- MMRV) = -1, 95% CI 2-sided [-2.4 to 0.8]

8. Secondary Outcome: Percentages of Subjects With hSBA ≥1:4 and hSBA ≥1:8 Following One Dose of MenACWY-CRM Vaccine
Description: The percentages of subjects with hSBA ≥1:4 and hSBA ≥1:8 after one dose of MenACWY-CRM vaccine (at 7-9 months), are reported
Time Frame: 1 month post vaccine dose 1
Population: The analysis was performed on the MenACWY per-protocol population
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY-CRM
Number analyzed (Participants) | 349
Percentages of subjects
  Serogroup A hSBA ≥1:4 | 63 [57 to 68]
  Serogroup A hSBA ≥1:8 | 50 [45 to 56]
  Serogroup C (N=199) hSBA ≥1:4 | 93 [88 to 96]
  Serogroup C (N=199) hSBA ≥1:8 | 88 [83 to 92]
  Serogroup W-135 (N=199) hSBA ≥1:4 | 48 [41 to 55]
  Serogroup W-135 (N=199) hSBA ≥1:8 | 37 [30 to 44]
  Serogroup Y (N=196) hSBA ≥1:4 | 41 [34 to 49]
  Serogroup Y (N=196) hSBA ≥1:8 | 31 [24 to 38]

9. Secondary Outcome: Geometric Mean Titers After One Dose of MenACWY-CRM Vaccine
Description: The immunogenicity of one dose of MenACWY-CRM vaccine given at 7 to 9 months of age was assessed in terms of GMTs directed against N.meningitidis serogroups A, C, W-135, and Y.
Time Frame: 1 month post vaccine dose 1
Population: The analysis was performed on the MenACWY per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM
Number analyzed (Participants) | 349
Titers
  Serogroup A | 8.16 [6.96 to 9.58]
  Serogroup C (N=199) | 26 [22 to 31]
  Serogroup W-135 (N=199) | 5.11 [4.15 to 6.29]
  Serogroup Y (N=196) | 4.09 [3.36 to 4.98]

10. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events After Vaccination
Description: Safety and tolerability of MenACWY-CRM and MMRV vaccines when given concomitantly compared to when either MenACWY-CRM or MMRV vaccine was administered alone is reported in terms of the number of subjects with local and systemic adverse events after vaccination.
  Systemic reactions including axillary temperature reported during 28 days after vaccination at 12 months of age. These included the following systemic reactions: Measles-like rash, Rubella-like rash, Varicellalike rash, injection site rash, Mumps-like symptoms and axillary temperature.
Time Frame: upto 7 days after any vaccination
Population: The analysis was performed on the safety set population
Measure: Number; unit: Participants
Arm/Group | MenACWY-CRM+MMRV | MenACWY-CRM | MMRV
Number analyzed (Participants) | 500 | 500 | 597
Participants
  Local Reactions | 278 | 298 | 316
  Injection(Inj.) site Tenderness [MenACWY-CRM] | 133 | 129 | 0
  Inj. site Erythema [MenACWY-CRM] | 153 | 159 | 0
  Inj.site Induration [ MenACWY-CRM] | 74 | 74 | 0
  Inj.site Tenderness [MMRV (N=455,424,592)] | 105 | 102 | 179
  Inj.site Erythema [MMRV (N=456,425,593)] | 156 | 145 | 224
  Inj. site Induration [MMRV (456,424,593)] | 90 | 60 | 102
  Systemic Reactions | 371 | 372 | 381
  Rash (N=500,499,595) | 54 | 44 | 46
  Change in eating habits (N=475,483,550) | 132 | 136 | 105
  Sleepiness (N=500,499,595) | 219 | 199 | 197
  Persistent crying (N=475,483,550) | 135 | 152 | 109
  Irritability (N=500,500,595) | 273 | 298 | 298
  Vomiting (N=500,499,595) | 66 | 74 | 36
  Diarrhea (N=500,499,595) | 120 | 123 | 107
  Fever ( N=499,500,596) | 58 | 78 | 42
  Other | 208 | 254 | 203
  Analgesic.Antipyr.Meds (N=499,499,594) | 208 | 254 | 203

11. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events After Vaccination
Description: The safety profile of MenACWY-CRM and MMRV vaccines when given concomitantly as compared to when MenACWY-CRM or MMRV was given alone is reported in terms of number of subjects reporting unsolicited adverse events (AEs), medically significant adverse events and serious adverse events (SAEs) after vaccination.
Time Frame: Day 1- Day 180 (Through out the study)
Population: This analysis was done on the safety set population
Measure: Number; unit: Participants
Arm/Group | MenACWY-CRM+ MMRV | MMRV | MenACWY-CRM
Number analyzed (Participants) | 500 | 597 | 500
Participants
  Any AE | 335 | 311 | 353
  At least probably related AEs | 70 | 2 | 63
  SAEs | 18 | 9 | 19

ADVERSE EVENTS:
Time Frame: All solicited adverse events (AEs) were collected upto Day 7 after each vaccination. All SAEs and unsolicited AEs were collected throughout the study (Day 1-Day 180).
Arm/Group | MenACWY-CRM+ MMRV | MMRV | MenACWY-CRM
Serious Adverse Events (participants affected / at risk) | 18/500 | 9/597 | 19/500
Other Adverse Events (participants affected / at risk) | 433/500 | 482/597 | 442/500
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACWY-CRM+ MMRV (N=500) | MMRV (N=597) | MenACWY-CRM (N=500)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Systemic inflamatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CROUP infectious (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 3 (3)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infections (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Toxic shock syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 3 (3)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Feeding disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tethered cord syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACWY-CRM+ MMRV (N=500) | MMRV (N=597) | MenACWY-CRM (N=500)
Diarrhoea (Gastrointestinal disorders) | 125 (125) | 114 (114) | 128 (128)
Teething (Gastrointestinal disorders) | 41 (41) | 41 (41) | 60 (60)
Vomiting (Gastrointestinal disorders) | 68 (68) | 43 (43) | 79 (79)
Injection site erythema (General disorders) | 219 (219) | 224 (224) | 230 (230)
Injection site induration (General disorders) | 128 (128) | 102 (102) | 115 (115)
Injection site pain (General disorders) | 163 (163) | 180 (180) | 188 (188)
Irritability (General disorders) | 273 (273) | 299 (299) | 299 (299)
Pyrexia (General disorders) | 90 (90) | 70 (70) | 114 (114)
Otitis media (Infections and infestations) | 92 (92) | 40 (40) | 120 (120)
Upper respiratory tract infection (Infections and infestations) | 71 (71) | 20 (20) | 92 (92)
Crying (Nervous system disorders) | 135 (135) | 109 (109) | 152 (152)
Somnolence (Nervous system disorders) | 219 (219) | 197 (197) | 199 (199)
Eating disorder (Psychiatric disorders) | 132 (132) | 105 (105) | 136 (136)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 26 (26) | 29 (29) | 30 (30)
Rash (Skin and subcutaneous tissue disorders) | 76 (76) | 87 (87) | 52 (52)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No